CLINICAL TRIAL: NCT02418403
Title: Consumer-directed Financial Incentives to Increase Advance Care Planning Among Medi-Cal Patients
Brief Title: Consumer Engagement to Increase Advance Care Planning: Patient Randomization
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Amber Barnato, MD, MPH, MS, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: PRO14110340
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Advance Care Planning

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PREPARE (Active Comparator): Access to "Prepare for Your Care" website and written encouragement to discuss ACP with one's PCP.
  Interventions: Behavioral: Educational website
- PREPARE+financial incentive (Experimental): Access to "Prepare for Your Care" website and written encouragement to discuss ACP with one's PCP; offer of $50 to complete the website and entry into $1000 lottery for discussing ACP with one's PCP.
  Interventions: Behavioral: Financial incentive; Behavioral: Educational website

INTERVENTIONS:
Behavioral: Financial incentive — Offer of money designed to overcome barriers to advance care planning.
  Arms: PREPARE+financial incentive
Behavioral: Educational website — Research-verson of the "Prepare for your care" website (www.prepareforyourcare.org)

SUMMARY:
This is a study of the effect of consumer-directed financial incentives on completion of advance care planning among Medi-Cal patients.

DETAILED DESCRIPTION:
Older adults receiving primary care from one of three clinics contracting with Partnership HealthPlan of California, a multi-county Medi-Cal managed care plan will be mass randomized to receiving educational materials regarding advance care planning with or without a financial reward for completing advance care planning.

ELIGIBILITY:
Inclusion Criteria:

* Partnership HealthPlan of California enrollee
* Receipt of primary care from one of 3 participating clinics (Ole, Petaluma, West County)
* Age > 65

Exclusion Criteria:

* > 75

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 376 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Having an advance care planning conversation with one's primary care provider | 3 months
  Primary care providers' documentation of an advance care planning conversation in the chart and/or via a Partnership HealthPlan of California ACP attestation form.

SECONDARY OUTCOMES:
Completion of "Prepare for Your Care" website modules | 3 months
  Logging into the website, completing the modules, and creating an action plan

CONTACTS AND LOCATIONS:
Overall Officials: Amber Barnato, MD MPH MS, Principal Investigator — University of Pittsburgh
Locations (1):
- Partnership HealthPlan of California, Fairfield, California, United States